CLINICAL TRIAL: NCT04180709
Title: Randomised Study of Web-based CBT Intervention (Sleepio) to Reduce Insomnia and Improve Social Recovery in Early Psychosis (CRISP)
Brief Title: CBT to Reduce Insomnia and Improve Social Recovery in Early Psychosis
Acronym: CRISP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Collaborators: Cambridgeshire and Peterborough NHS Foundation Trust (Other); Cambridge Cognition Ltd (Industry); Big Health Inc. (Industry)
Responsible Party: Principal Investigator, Peter Jones, Professor of Psychiatry / Deputy Head of Clinical School, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: M00915; RNAG-521 (Other Grant/Funding Number: Cambridgeshire and Peterborough NHS Foundation Trust (CPFT)); 224101 (Other: Integrated Research Application System (IRAS)); 19/EE/0352 (Other: NHS HRA - Cambridge South Research Ethics Committee)
Record Dates: First submitted 2019-10-28; First posted 2019-11-27 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Psychotic Disorders; Psychosis; Sleep
Keywords: Cognition; Social Recovery; Immunopsychiatry; Daily function; Sleep disturbances; Insomnia
MeSH Terms: conditions — Psychotic Disorders; Parasomnias; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: This is a randomised parallel study design, with five points of measurements. Participants will receive either the Sleepio online intervention + treatment as usual (TAU) or TAU alone over an 8-week period. A follow-up period will be conducted for an additional 8 weeks. The original TAU group will be offered the intervention during this period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleepio Intervention + Treatment As Usual (TAU) (Experimental): Participants will receive the online Sleepio intervention to be completed approximately once per week, at least 6 sessions during the 8-week period, and complete daily sleep diaries. In addition they will continue their treatment as usual (TAU) with the CAMEO Early Intervention in Psychosis CPFT or Early Intervention in Psychosis Services NSFT care team.
  Interventions: Device: Sleepio
- Treatment As Usual (TAU) alone (No Intervention): Participants will continue their treatment as usual (TAU) with their Early Intervention in Psychosis care team. They will however be offered access to the Sleepio intervention during the follow-up period of the study.

INTERVENTIONS:
Device: Sleepio — Sleepio is an online cognitive behavioural therapy (CBT) based intervention designed to treat insomnia, conducted is 6 sessions. The program is an automated media-rich web-based application that is driven dynamically by baseline, adherence, performance and progress data. At the beginning of each session The Prof conducts a progressive review with the participant exploring the diary data submitted the week prior that includes sleep status and pattern, as well as progress based on goals previously set by the participant. The information, support and advice are personally tailored based on underlying algorithms.
  Arms: Sleepio Intervention + Treatment As Usual (TAU)

SUMMARY:
Sleep disturbances and cognitive dysfunction are consistently reported as extremely troublesome aspects of psychotic illnesses. While sleep disturbances are not included in definitions of psychosis they are associated with poor levels of daily function and impaired social recovery. Despite sleep problems being documented as co-occurring with psychosis, sleep remains unexamined as a potential therapeutic target pathway for social recovery. Specific areas of cognition are known to be associated with psychosis, sleep deficits and daily function, yet these have not been tested as possible mediators of the association between improved sleep and better daily function and social recovery.

This study will examine the relationship between sleep quality, daily function and ultimately social recovery in early psychosis. A secondary aim will examine whether specified areas of cognition (i.e. attention, memory, executive function, social and emotional recognition) mediate the proposed association between sleep and social recovery. Participants will have experienced a first episode psychosis and be currently engaged with CAMEO early intervention, in Cambridgeshire and Peterborough NHS Foundation Trust (CPFT) or Early Intervention in Psychosis Services (EIS), in Norfolk and Suffolk NHS Foundation Trust (NSFT). Cameo CPFT and Early Intervention in Psychosis Services NSFT are services for people aged 14-65 years old who are experiencing symptoms of psychosis for the first time (http://www.cameo.nhs.uk and https://www.nsft.nhs.uk/adults/service/early-intervention-in-psychosis-services-norfolk-and-waveney-103/). A publicly available, online intervention based on cognitive behavioural therapy (CBT) for insomnia (Sleepio) will be utilised to improve sleep. Participants will be randomised to receive the intervention + treatment as usual (TAU) through their early intervention team or TAU alone over an eight-week period. The entire study will last for seventeen weeks including an eight-week follow-up period.

DETAILED DESCRIPTION:
The study will take place in three stages; an initial survey, an eight week study period and a follow-up period for an additional eight weeks.

Stage One: Perceptions of Sleep Problems and Their Treatment in Psychosis:

Clinicians and service users will receive an online link to a short 18-question survey (primarily multiple choice) that should take approximately 5 min to complete. Although they can complete this online, a paper copy can be provided if they prefer to handwrite their answers.

Stage Two: Randomised 8 Week Study:

At our initial phone or NHS approved video platform meeting participants will be invited to ask any questions they have. If they choose to participate in our study, they will be asked to read and sign a consent form virtually or through the post. They will also be asked their preferred method of contact during the study so that the primary researcher can arrange appointments and check in once or twice per week. This will allow them to ask any questions which may arise and offer assistance if they are having any challenges with logging in or participation. They will also be informed that they have the right to withdraw from the study at any point and this will have no affect on their ongoing treatment through the EIS they are currently supported by.

Following consent to take part in the research study participants will answer some screening questions and complete a short 8-question assessment (about 5-10 min). Participants will be asked general questions about themselves and with their consent some diagnostic information will be obtained from clinical records. Following this they will be randomly assigned to one of two groups. The first will utilise the Sleepio intervention during the 8-week study period, along with their usual treatment from the EIS team and the second group will just continue their usual treatment for this 8-week period.

Prior to starting the study period, we will ask participants to monitor their sleep for one week using a nightly sleep diary (2-3 minutes) and by asking them to wear an actigraphy watch, a small device that records movement, light and near body temperature. At the end of this week we will complete baseline assessments with all participants and provide them with access logins for Sleepio. Most of these can be completed online and should only take about 35 minutes. The Guided Web-Based CANTAB cognitive tests will take approximately 25 min, be done online with video support from the researcher, and will include breaks for participant comfort. They will also have the option of completing some or all of the self assessments over the phone, video call or by post if they prefer.

The researcher administered assessments will be done with Camice Revier, the lead researcher, and should take around 15 min.

During the 8-week intervention period participants will complete weekly online 20-30 minute interventions via Sleepio (6 interventions in total, as occasional delays are accommodated for and expected) and complete nightly sleep diaries online via Sleepio (2-3 minutes).

After 4-weeks of the study participants will be asked to do a second round of assessments. This round has fewer measures and should only take about 20 minutes for the online assessments, 25 minutes for the Guided CANTAB cognitive tests and around 10 minutes for those done over the phone or video meeting.

During week 7 of the study we'll ask participants to again wear the actigraphy watch for another week.

The third round of assessments will take place at the end of the 8-week study period and will be the same duration as the original assessments: online about 35 min, CANTAB cognitive tests about 25 min and over the phone or video meeting about 10 min.

Stage Three: Follow-up and Anonymous Feedback Questionnaire:

During the follow-up period we will invite those who were not randomised into the treatment group to utilise the Sleepio intervention at this time.

All of the assessments will take place in the same order and duration as they did during the initial study period.

During week 7 of the follow-up period we'll ask participants, one final time, to complete the sleep diaries and wear the actigraphy watch for a final week.

Following the study participants will be invited to complete an anonymous feedback questionnaire. This is intended to provide a way for them to communicate any input or suggestions based on their experience and to help us improve the way we do things.

They will be offered the option of researchers contacting them for additional follow-up or to be invited to participate in related studies. There is no obligation for them to do so and they can indicate on their consent form whether they are willing to be contacted at a later date (within 5 years).

ELIGIBILITY:
Inclusion Criteria:

* Experiencing or having experienced a First Episode of Psychosis (FEP) within the past 5 years.
* Currently participating in CPFT CAMEO EIPS or NSFT EIS and intending to continue TAU with the specified service for at least the next 4 months.
* Mental capacity for consent.
* Currently experiencing threshold level (score ≤ 16 on SCI-8) of disrupted sleep.
* Adults 18 years or older.
* Ability to understand and follow therapeutic instructions necessary for experiment and respond to online questionnaires.
* Illness duration less than or equal to 5 years. Onset of illness was defined as first contact with psychiatric services for psychotic symptoms.
* Access to the internet.

Exclusion Criteria:

* Too unwell to viably participate in study.
* A diagnosis of drug induced psychosis or bipolar disorder.
* Psychotic disorder due to a medical or physical disease (i.e. considered to have an organic basis).
* Current drug or alcohol dependency.
* Currently taking prescribed sleep medication or intending to do so during study.
* Currently doing night shift work.
* Travel over 2 time zones during or within two weeks prior to assessment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Work and Social Adjustment Scale (WSAS) score at week 9 of study | Measure completed at baseline (start of week 1) and week 9.
  WSAS is a simple and reliable measure of impaired functioning. Scores range from 0-40, with lower scores representing better functioning, scores 0-10 are considered subclinical, 11-20 associated with significant functional impairment but less severe clinical symptomology, and >20 suggest moderately severe functional impairment (Mundt et al. 2002).

SECONDARY OUTCOMES:
Time Use Survey - Structured Hours (TUS-SH) | Measure completed in weeks 1, 5, 9, 13 and 17.
  Social recovery will be measured using an adapted versions of the Time Use Survey (TUS) Structured Hours, which has been previously validated for use as a social recovery measure by Hodgekins, Fowler and colleagues, and utilised in the National EDEN study (Hodgekins et al. 2015; Hodgekins 2012; Fowler et al. 2009). This will be adapted to a reduced interview to include only those areas relevant to the social recovery measure, hence the Time Use Survey-Structured Hours (TUS-SH).
Patient Health Questionnaire (PHQ-9) | Measure completed in weeks 1, 5, 9, 13 and 17.
  PHQ-9 is a self-administered measure of depression, which scores all 9 of the DSM-IV criteria for depression. Scores range from 0-27, with 5-9 indicating minimal symptoms, 10-14 minor depression, 15-19 moderately severe major depression and ≥20 severe major depression.
Rapid Visual Information Processing (RVP) / CANTAB Cognitive Test | Measure completed in weeks 1, 5, 9, 13 and 17.
  iPad delivered cognitive test of sustained attention.
Paired Associates Learning (PAL) / CANTAB Cognitive Test | Measure completed in weeks 1, 5, 9, 13 and 17.
  iPad delivered cognitive test of visual episodic memory.
Spatial Working Memory (SWM) / CANTAB Cognitive Test | Measure completed in weeks 1, 5, 9, 13 and 17.
  iPad delivered cognitive test of working memory and strategy.
Emotion Recognition Task (ERT) / CANTAB Cognitive Test | Measure completed in weeks 1, 5, 9, 13 and 17.
  iPad delivered cognitive test of emotional recognition.
Global Assessment of Functioning (GAF) (split version / subscales GAF-D & GAF-S) | Measure completed in weeks 1, 9 and 17.
  GAF is an assessment of psychological, social and occupational functioning along a hypothetical continuum of mental health/illness. It is suggested that symptom scale for degree of severity be considered to cover the past 3 days prior to assessment but time frames can be varied based on the intention of use (Aas 2011). However by utilising the split version of this measure, the symptom and function scores can be evaluated and considered independently. This has been shown to be highly consistent across experienced raters, so sufficient training and utilisation may be fundamental to its efficacy (Pedersen et al. 2007). Scores range from 0-100 with higher scores representing better functioning across symptomatic and functional domains (Hall 1995).
Change from baseline Work and Social Adjustment Scale (WSAS) score at week 17 | Measure completed at baseline (start of week 1) and week 17.
  WSAS is a simple and reliable measure of impaired functioning. Scores range from 0-40, with lower scores representing better functioning, scores 0-10 are considered subclinical, 11-20 associated with significant functional impairment but less severe clinical symptomology, and >20 suggest moderately severe functional impairment (Mundt et al. 2002).
Change from baseline Work and Social Adjustment Scale (WSAS) score at week 5, to correct for confounding in mediation analysis | Measure completed at baseline (start of week 1) and week 5.
  WSAS is a simple and reliable measure of impaired functioning. Scores range from 0-40, with lower scores representing better functioning, scores 0-10 are considered subclinical, 11-20 associated with significant functional impairment but less severe clinical symptomology, and >20 suggest moderately severe functional impairment (Mundt et al. 2002).
Change from baseline Work and Social Adjustment Scale (WSAS) score at week 13, to correct for confounding in mediation analysis | Measure completed at baseline (start of week 1) and week 13.
  WSAS is a simple and reliable measure of impaired functioning. Scores range from 0-40, with lower scores representing better functioning, scores 0-10 are considered subclinical, 11-20 associated with significant functional impairment but less severe clinical symptomology, and >20 suggest moderately severe functional impairment (Mundt et al. 2002).

OTHER OUTCOMES:
Sleep Condition Indicator (SCI-8) | Measure completed in weeks 1, 5, 9, 13 and 17.
  SCI-8 this measure is validated against DSM-5 criteria for insomnia, including sleep quality and daytime function over the previous week. It is utilised within the Sleepio intervention and was the primary outcome measure for the OASIS randomised controlled trial (Freeman et al. 2017). This eight-item assessment questionnaire includes: 'concerns about getting to sleep, remaining asleep, sleep quality, daytime functioning, daytime performance, duration of sleep problem, nights per week having a sleep problem and extent troubled by poor sleep'(Espie, Kyle, Hames, et al. 2014). It has a robust internal consistency (α≥0.86) and showed convergent validity with the Pittsburgh Sleep Quality Index (PSQI) and Insomnia Severity Index (ISI) (Espie, Kyle, Hames, et al. 2014). Scores range from 0-32 with higher scores indicating better sleep, scores below 17 identifying insomnia in 89% of cases (Espie, Kyle, Hames, et al. 2014; Freeman et al. 2017).
Insomnia Severity Index (ISI) | Measure completed in weeks 1, 9 and 17.
  ISI is a measure specifically designed as a brief self-administered measure of insomnia and outcomes for use in their treatment within research. It corresponds to the DSM-IV criteria for insomnia and measures perception and severity of symptoms within the previous 2 weeks. Scores range from 0-28, 0-7 indicating no significant insomnia, 8-14 sub threshold insomnia, 15-21 moderate clinical insomnia, and 22-28 severe clinical insomnia (Smith & Wegener 2003; Bastien et al. 2001). It has been validated as a web-based measure with internal consistency of ≥88% (Thorndike et al. 2011).
Pittsburgh Sleep Quality Index (PSQI) | Measure completed in weeks 1, 9 and 17.
  PSQI is a self-report 19-item measure that retrospectively measures sleep quality and disturbances over the previous month. The domains of sleep quality included are: sleep wake patterns, duration of sleep, sleep latency, the frequency and severity of specific sleep-related problems and impact on daytime function. Scores range from 0-21, with higher scores indicating poorer sleep quality. The empirically derived cut-off score is >5 to distinguish poor sleepers with severe difficulties in at least 2 domains, or moderate difficulties in more than 3 domains. This cut-off correctly identifies 88.5% of patients, with a sensitivity of 89.6% and specificity of 86.5% (Buysse et al. 1989; Smith & Wegener 2003).
Validation of Sleep Diaries by comparison with actigraphy activity data | Monitoring will be done for a complete week just prior to week 1, during week 8 and 16. Sleep diaries are collected nightly during this same period.
  Nightly sleep diaries will be reported online using the Sleepio.com online diary.
  GENEActive actigraphy watch will collect raw data of activity. Which will record sleep patterns objectively. This will be compared with sleep diaries for consistency of subjective measure with objective measure.
  The actigraphy data will be considered for L5 (lowest 5 hours of activity) M10 (highest 10 hours of activity) and relative amplitude (ratio between L5 and M10). This will then be compared with the nightly sleep diaries for the same period to determine percentage of consistency of reporting.
COVID-19 Brief Questionnaire (COVID-19-B) | Measure completed in weeks 1, 5, 9, 13 and 17.
  This is a short 7 question (3 minute) survey to allow us to collect basic data on the impact of the ongoing pandemic on participants.

CONTACTS AND LOCATIONS:
Overall Officials: Peter B Jones, PhD MD, Principal Investigator — University of Cambridge
Locations (1):
- Cameo Early Intervention, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No